CLINICAL TRIAL: NCT04744714
Title: Establishment of Gestational Weight Gain Criteria for Pregnant Women With Gestational Diabetes Mellitus in China: a Multicenter Prospective Cohort Study
Brief Title: Gestational Weight Gain Criteria for Pregnant Women With Gestational Diabetes Mellitus in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: GWG2021
Record Dates: First submitted 2021-01-27; First posted 2021-02-09 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Gestational Weight Gain
Keywords: gestational weight gain; gestational diabetes mellitus
MeSH Terms: conditions — Gestational Weight Gain; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, urine, tissue (placenta and umbilical cord)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GDM group: questionnaire survey and clinical follow-up
- non-GDM group: questionnaire survey and clinical follow-up

SUMMARY:
Appropriate gestational weight gain (GWG) is a key factor in balancing maternal and neonatal needs of nourishment and health, which is especially important in women with gestational diabetes mellitus (GDM). However, there are no specific guidelines for GWG in Chinese pregnant women and even for GDM pregnant women.This project intends to fill in the gaps of this field through multi-center large sample prospective cohort study.

DETAILED DESCRIPTION:
Inappropriate gestational weight gain (GWG) is an important risk factor affecting adverse pregnancy outcomes. However, the current guidelines for GWG are based on American population and may not apply to pregnant women in China, especially for those with gestational diabetes mellitus (GDM) who have high risk factors. The big gaps in academic-related fields need to be filled.

Our research group has previously found the heterogeneous relationships between GWG and adverse outcomes in GDM women with different abnormal glucose metabolism. Therefore, based on the principles of precision medicine, this project intends to establish for the first time the GWG standard for Chinese pregnant women to optimize the GWG management through a multicenter prospective cohort study. At the same time, specific GWG guidelines applicable to GDM women with different glucose metabolism abnormalities were innovatively constructed. Our study will provide strong evidence for stratified management and precise intervention of GDM pregnant women, which is of great significance to ensure health of both mothers and their offspring.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age: 20-49 years;
* Natural conception;
* Single pregnancy;
* Plan to have routine prenatal examinations and give birth in the research center;
* No plan to move within two years;
* No second pregnancy within two years;
* Willing to cooperate with the hospital to follow up after childbirth.

Exclusion Criteria:

* Have diseases that affect metabolic function or even threaten the life of the mother and fetus before pregnancy, such as diabetes, hypertension, heart disease, liver and kidney diseases, thyroid diseases, autoimmune diseases, malignant tumors, AIDS, etc.;
* Assisted reproduction;
* Multiple pregnancy;
* Fetus has a known deformity or genetic defects;
* Incomplete clinical data.

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This project intends to recruit pregnant women who go to the research center for routine prenatal examination and OGTT screening.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal outcomes | Through delivery completion, up to 40 weeks
  Including pregnancy-induced hypertension, preterm delivery, abortion, delivery way and so on. They are diagnosed by clinicians and the data is gathered from medical records.
Neonatal outcomes | Through delivery completion, up to 40 weeks
  Birth weight（in gram), birth height (in centimetre), gestational week (in week) and so on. They are diagnosed by clinicians and the data is gathered from medical records.

SECONDARY OUTCOMES:
glucose metabolism index | postpartum 42 days
  OGTT results (mmol/L), HbA1c (%) and so on
offspring | postpartum 42 days
  weight (in gram), height (in centimetre), feeding situation (breast feeding or artificial feeding) and so on.
annual follow-up results | 1 or 2 years after delivery
  Annual questionnaire and physical examination, including weight (in kilogram), height (in metre), disease history, diet surveys and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoxia Liang, M.D., Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital School of Medicine Zhejiang University, Hangzhou, China